CLINICAL TRIAL: NCT05521282
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Qianglidingxuan Tablets in the Treatment of Mild to Moderate Essential Hypertension With Hyperactivity of Liver Yang
Brief Title: The Efficacy of Qianglidingxuan Tablets in the Treatment of Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine (Unknown); Jilin Provincial Hospital of Traditional Chinese Medicine, Affiliated Hospital of Changchun University of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, kuiwu Yao, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QLDXP-202002
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Medicine, Chinese Traditional
Keywords: Hypertension; Qianglidingxuan tablet; Traditional Chinese medicine; Randomized controlled trial; Chinese patent medicine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Based on the basic treatment, Qianglidingxuan Tablets were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.
Who Masked: Participant
Masking Description: Based on basic treatment, Qianglidingxuan mimetics were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Based on the basic treatment, Qianglidingxuan Tablets were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.
  Qianglidingxuan Tablets:
  Specifications: 60 tablets per bottle; Storage: airtight, moisture-proof; Active ingredients:Gastrodia elata, Eucommia ulmoides, wild chrysanthemum, Eucommia ulmoides leaves, Chuanxiong; Manufacturer: Shaanxi Hanwang Pharmaceutical Co., LTD.
  Interventions: Drug: Treatment group
- Control group (Placebo Comparator): Based on basic treatment, Qianglidingxuan Tablets mimetics were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.
  Qianglidingxuan Tablets mimetics:
  Specifications: 60 tablets per bottle; Storage: airtight, moisture-proof; Active ingredients:NA; Manufacturer: Shaanxi Hanwang Pharmaceutical Co., LTD.
  Interventions: Drug: Treatment group

INTERVENTIONS:
Drug: Treatment group — Based on the basic treatment, Qianglidingxuan Tablets were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.

SUMMARY:
Research purpose: This study was a multicenter, randomized, double-blind, placebo-controlled, post-marketing clinical study in Chinese patients with essential hypertension to evaluate the efficacy and safety of Qianglidingxuan tablets(QLT) in the treatment of blood pressure in patients with mild to moderate essential hypertension.

1. Subject:

   Patients diagnosed as essential hypertension with clinical grade 1-2.
2. Interventions:

   ①Basic treatment plan:Patients in both groups were required to have a low-salt, low-fat diet, quit smoking, limit alcohol, eat more vegetables, moderate exercise, control body weight, and amlodipine besylate tablets (5mg, QD).

   ②Treatment group: Based on the basic treatment, QLT was given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.

   ③Control group: Based on basic treatment, QLT mimetic were given 6 tablets/time, 3 times a day, and warm water was given for 12 weeks.
3. Treatment and follow-up cycle:

   Patients in both groups were treated for 12 weeks and followed up to the end of 48th week after treatment.
4. Provisions of concurrent treatment:

   Any combined treatment used during the study should be recorded in the CRF, including drug name (generic name/trade name), starting time, administration dose, method of administration, termination time, indication, etc
5. Efficacy evaluation:

   ①Primary outcome measure: the change from baseline in office blood pressure after 12 weeks of treatment.

   ②Secondary efficacy indicators: 24-hour ambulatory blood pressure, heart rate, blood lipids, homocysteine, CRP, baPWV. TCM syndromes (including vertigo, headache, impatience and irritability, red face, red eyes, dry mouth, bitter mouth, tinnitus, insomnia, multiple dreams, constipation, urination, etc.)

   ③Safety indicators: adverse events, vital signs, physical examination, laboratory examination
6. Statistics:

SAS® 9.4 was used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75 years.
2. Patients diagnosed as essential hypertension with clinical grade 1-2.
3. Diagnosis of hyperactivity of liver Yang upper syndrome by TCM syndrome differentiation.
4. Patients signed the informed consent with good compliance and could cooperate with the follow-up and review.

Exclusion Criteria:

1. Secondary hypertension: renal hypertension (renovascular hypertension, renal parenchymal hypertension), pheochromocytoma, primary aldosteronism, Cushing syndrome, abdominal aortic coarctation, etc.
2. Coronary atherosclerotic heart disease, acute attack of chronic heart failure, malignant arrhythmia, valvular heart disease, cardiomyopathy and other serious cardiovascular diseases.
3. Acute cerebrovascular diseases such as cerebral infarction and cerebral hemorrhage.
4. Severe psychological disorder, intellectual disability or language disorder, resulting in inability to fully cooperate with the study and inability to complete the study.
5. Any laboratory test index before screening met the following criteria: admission liver and kidney function indicated that ALT, AST > 1.5 times the upper limit of normal value, Cr > 1.2 times the upper limit of normal value (refer to the laboratory normal range of the research center); Other clinically significant laboratory abnormalities that were deemed unsuitable for enrollment by the investigator.
6. Allergic constitution or allergic to strong fixed glare tablets, excipients or similar ingredients of the trial drug.
7. Suspected or with a history of alcohol or drug abuse.
8. Pregnant, lactating women or those who plan to get pregnant recently or are unwilling to use contraceptive measures;.
9. Patients who had participated in other clinical trials within 3 months before enrollment.
10. Patients deemed by the investigator to be ineligible for enrollment in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Clinic blood pressure | Baseline, month 4, month 12
  Changes in systolic and diastolic blood pressure from baseline to follow up

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure | Baseline, month 4, month 12
  Changes in daytime systolic BP, daytime diastolic blood pressure, nighttime systolic blood pressure, nighttime diastolic blood pressure, 24h mean systolic blood pressure, and 24h mean diastolic blood pressure from baseline to follow up
Heart rate | Baseline, month 4, month 12
  Changes in heart rate from baseline to follow up
Blood lipids | Baseline, month 4, month 12
  Changes in blood lipids（triglyceride, total cholesterol, low-density lipoprotein cholesterol, and high-density lipoprotein cholesterol）from baseline to follow up
BMI | Baseline, month 4, month 12
  Changes in BMI from baseline to follow up
Homocysteine | Baseline, month 4, month 12
  Changes in homocysteine from baseline to follow up
C reactive protein | Baseline, month 4, month 12
  Changes in C reactive protein from baseline to follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin J, Wang Q, Zhong D, Zhang J, Yuan T, Wu H, Li B, Li S, Xie X, An D, Deng Y, Xian S, Xiong X, Yao K. Efficacy and safety of Qiangli Dingxuan tablet combined with amlodipine besylate for essential hypertension: a randomized, double-blind, placebo-controlled, parallel-group, multicenter trial. Front Pharmacol. 2023 Jul 10;14:1225529. doi: 10.3389/fphar.2023.1225529. eCollection 2023. PMID 37492087